CLINICAL TRIAL: NCT04722458
Title: Turkish Validity and Reliability of LURN SI-29 Questionnaire Form in Patients With Lower Urinary Tract Symptoms
Brief Title: Turkish Validation and Reliability of LURN SI-29 Questionnaire in Patients With Lower Urinary Tract Symptoms
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ahmet Tahra, Assistant Professor of Urology, Istanbul Medeniyet University
Other Study IDs: 2021-0028
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Lower Urinary Tract Symptoms; Urinary Incontinence
Keywords: Lower urinary tract symptoms; Patient reported outcomes; Questionnaire
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Lower urinary tract sypmtoms: Patients with Lower urinary tract sypmtoms over 18 years old will be included to this study
  Interventions: Other: Lower Urinary Tract Dysfunction Research Network Symptom Index-29 (LURN SI-29); Other: IPSS; Other: UDI-6

INTERVENTIONS:
Other: Lower Urinary Tract Dysfunction Research Network Symptom Index-29 (LURN SI-29) — LURN SI-29
Other: IPSS — International Prostate Symptom Score
Other: UDI-6 — Urogenital Distress Inventory

SUMMARY:
Lower urinary tract symptoms is quite frequent in men and women. To better understand the the symptoms that characterize lower urinary tract, the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) has established the Symptoms of Lower Urinary Tract Dysfunction Research Network (LURN). In this study we aim to validate the LURN-29 score to Turkish language

ELIGIBILITY:
Inclusion Criteria:

* Patients with lower urinary tract symptoms, Over 18 years old,Patient with the cognitive ability to read

Exclusion Criteria:

* Patients above 18 years old

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with lower urinary tract symptoms over 18 will be included
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
LURN SI-29 Questionnaire | 3 months
  The subscale and total scores for the LURN SI-29 are normalized to a scale from 0 - 100
International Prostate Symptom Score-IPSS | 3 months
  The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
UROGENITAL DISTRESS INVENTORY- 6 | 3 months
  UDI-6 a six item symptom inventory, specific to symptoms associated with lower urinary tract dysfunction,and combines information on irritative, stress and obstructive/discomfort symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cella D, Smith AR, Griffith JW, Flynn KE, Bradley CS, Gillespie BW, Kirkali Z, Talaty P, Jelovsek JE, Helfand BT, Weinfurt KP; LURN Study Group. A new outcome measure for LUTS: Symptoms of Lower Urinary Tract Dysfunction Research Network Symptom Index-29 (LURN SI-29) questionnaire. Neurourol Urodyn. 2019 Aug;38(6):1751-1759. doi: 10.1002/nau.24067. Epub 2019 Jun 21. PMID 31225927
- [Result] Cella D, Smith AR, Griffith JW, Kirkali Z, Flynn KE, Bradley CS, Jelovsek JE, Gillespie BW, Helfand BT, Talaty P, Weinfurt KP; LURN Study Group. A New Brief Clinical Assessment of Lower Urinary Tract Symptoms for Women and Men: LURN SI-10. J Urol. 2020 Jan;203(1):164-170. doi: 10.1097/JU.0000000000000465. Epub 2019 Jul 31. PMID 31364922